CLINICAL TRIAL: NCT00033033
Title: Phase 2, Double-Blind, Placebo-Controlled Trial of Reserpine for the Treatment of Cocaine Dependence
Brief Title: Reserpine for the Treatment of Cocaine Dependence - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Cincinnati VA Medical Center (U.S. Federal Agency)
Responsible Party: Liza Gorgon / Clinical Trials Specialist, NIDA
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIDA-CTO-0001-1; NCT00024869 (obsolete NCT alias)
Record Dates: First submitted 2002-04-05; First posted 2002-04-08 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-08

CONDITIONS: Cocaine-Related Disorders; Substance-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders | interventions — Reserpine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Reserpine

SUMMARY:
The purpose of this study is to assess the efficacy and safety of reserpine for the treatment of cocaine dependence.

DETAILED DESCRIPTION:
To assess the efficacy and safety of reserpine in reducing cocaine use in subjects with cocaine dependence. This is a double-blind, placebo-controlled, parallel-group design with a 2 week baseline period.

ELIGIBILITY:
Inclusion Criteria:

Be at least 18 yrs of age; DSM-4 diagnosis of cocaine dependence; treatment seeking individuals; have the ability to understand and provide written informed consent; females of child bearing potential using appropriate birth control method

Exclusion Criteria:

Additional criteria available during screening at the site.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140
Dates: Start 2001-07; Study Completion 2003-05

PRIMARY OUTCOMES:
Cocaine use
Addiction severity
Cocaine withdrawal
Adverse events
Clinical improvement

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Somoza, M.D., Ph.D., Principal Investigator — Cincinnati VA Medical Center
Locations (3):
- United States (3):
  - Boston University Medical Center, Boston, Massachusetts
  - Cincinnati VA Medical Center, Cincinnati, Ohio
  - Dayton VA Medical Center, Dayton, Ohio

REFERENCES:
- [Derived] Winhusen TM, Lewis DF, Somoza EC, Horn P. Pharmacodynamics must inform statistics: an example from a cocaine dependence pharmacotherapy trial. ISRN Addict. 2014 Feb 5;2014:927290. doi: 10.1155/2014/927290. eCollection 2014. PMID 25969833
- [Derived] Winhusen TM, Somoza EC, Lewis DF, Kropp F, Theobald J, Elkashef A. An Evaluation of Substance Abuse Treatment and HIV Education on Safe Sex Practices in Cocaine Dependent Individuals. ISRN Addict. 2014 Mar 4;2014:912863. doi: 10.1155/2014/912863. eCollection 2014. PMID 25938124